CLINICAL TRIAL: NCT06222853
Title: A Clinical Study on the Safety and Efficacy of Chimeric Antigen Receptor T Cell Injection Targeting CD19 Gene in the Treatment of Refractory Systemic Lupus Erythematosus
Brief Title: Study of Therapeutic Efficacy of Anti-CD19 CAR-T Cells in Refractory Systemic Lupus Erythematosus
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Mao Jianhua, Professor, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEAM
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus; CAR-T Cell Therapy
Keywords: Systemic Lupus Erythematosus; CAR-T
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment group (Experimental): This is an open-label, single-arm, multicenter, investigator-initiated study. The study will primarily evaluate the Target Dose of 1×10^5 CAR+ cells/kg. The majority of subjects will be enrolled at this level to characterize efficacy and safety. Two exploratory dose levels-Low Dose (0.3×10^5 CAR+ cells/kg) and High Dose (3×10^5 CAR+ cells/kg)-are reserved for dose modification based on safety signals or preliminary efficacy data.
  Interventions: Biological: anti-CD19-CAR-T cells

INTERVENTIONS:
Biological: anti-CD19-CAR-T cells — The study will primarily evaluate the Target Dose of 1×10^5 CAR+ cells/kg. The majority of subjects will be enrolled at this level to characterize efficacy and safety.
  Two exploratory dose levels-Low Dose (0.3×10^5CAR+ cells/kg) and High Dose (3×10^5 CAR+ cells/kg)-are reserved for dose modification based on safety signals or preliminary efficacy data.

SUMMARY:
This is an investigator-initiated trial aimed at assessing the safety of anti-CD19 CAR-T cells in the treatment of refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a serious autoimmune disease that can lead to extensive damage in multiple organs and systems, ultimately resulting in disability and even death. Children with SLE are particularly at risk of organ damage, especially to the kidneys, and tend to have a more severe and protracted course of the disease compared to adults.

Currently, the primary treatment for SLE relies on glucocorticoids and immunosuppressants to alleviate symptoms. However, due to the absence of a curative treatment, patients often require lifelong medication. In recent years, biological agents such as belimumab and rituximab have been introduced for the treatment of SLE, but these agents cannot completely eliminate autoimmune B cells in the bone marrow, leading to unsatisfactory overall outcomes. Furthermore, stopping the drugs can lead to relapse, and there is still no cure for SLE, leaving patients facing the challenges of lifelong medication and an incurable disease.

Since 2019, CAR-T cell therapy has been successfully applied to autoimmune diseases. Clinical studies have demonstrated that targeted CD19 CAR-T cells hold significant therapeutic potential for SLE. These cells effectively slow down the pathological progression of SLE and can also effectively treat severe cases. Furthermore, targeted CD19 CAR-T cells are also expected to restore the immune system in SLE patients, potentially allowing them to discontinue lifelong medication and avoid serious long-term side effects of drugs like hormones and immunosuppressants. The purpose of this study is to assess the safety and efficacy of the anti-CD19 CAR-T cells in the treatment of refractory SLE.

ELIGIBILITY:
Inclusion Criteria

1. Age: ≥5 years old.
2. Refractory SLE Diagnosis:

   1. Diagnosed with SLE according to the 2019 EULAR/ACR classification criteria.
   2. Exhibit persistent moderate to severe disease activity (defined as a SLEDAI-2K score ≥ 8).
   3. Demonstrated failure or to achieve target disease control (LLDAS or remission) after a minimum of 6 months of standard-of-care therapy, including: high doses of glucocorticoids (≥1mg/kg/day prednisone or equivalent), hydroxychloroquine, and at least two DMARDs (including cyclophosphamide, MMF, azathioprine, methotrexate, cyclosporine, tacrolimus, sirolimus, leflunomide, tocilizumab, belimumab, and rituximab) for at least 6 months; or intolerant to conventional treatments.

   Note: Patients may also be eligible if they are documented as intolerant to these conventional treatments.
3. Disease Severity Validation: To ensure a "refractory" status, patients must satisfy at least one of the following:

   1. Active Major Organ Involvement (e.g., biopsy-proven Lupus Nephritis Class III, IV, or V; CNS lupus; or refractory hematological cytopenias).
   2. Steroid Dependence: Inability to taper glucocorticoid dose below 0.5 mg/kg/day (or equivalent) without a disease flare.
4. Organ Function:

   1. Cardiac: LVEF ≥ 55 %, with no significant clinical abnormalities on ECG.
   2. Renal: Estimated glomerular filtration rate (eGFR) 30 mL/min/1.73m2.
   3. Liver: AST and ALT ≤ 3.0 ULN, and total bilirubin ≤ 2.0 ULN.
   4. Pulmonary: No severe lung disease, with oxygen saturation (SpO2) ≥ 92% on room air.
5. Apheresis Suitability: Must meet institutional criteria for leukapheresis and have no contraindications to peripheral blood mononuclear cell (PBMC) collection.
6. Contraception: Females of childbearing age must have a negative urine pregnancy test at screening and agree to use effective contraceptive measures from enrollment until 1 year after MC-1-50 cell infusion.
7. Informed Consent: Voluntary written informed consent must be obtained from the subject (if applicable) and their lawful guardians prior to any screening procedures.

Exclusion Criteria:

1. Prior Cell Therapy: Previous treatment with any CAR-T cell therapy or other genetically modified effector cell products.
2. Neurological/CNS Involvement:

   1. Active central nervous system (CNS) lupus requiring clinical intervention within 60 days of screening (including seizures, delirium, or cerebrovascular events).
   2. Evidence of significant structural CNS damage on MRI or a history of severe seizures that may lower the threshold for ICANS.
3. Severe Renal Impairment and Fibrosis:

   1. Receiving renal replacement therapy (dialysis) within 3 months prior to infusion.
   2. Irreversible Renal Damage: Documented high chronicity on baseline biopsy (e.g., Chronicity Index >6/12) or extensive renal fibrosis, as these patients are unlikely to achieve functional recovery despite immunological remission.
   3. Significant nephropathy likely requiring high-dose glucocorticoids (≥1mg/kg/day prednisone or equivalent) or intensified DMARDs within 3 months of infusion.
4. Cardiac Conditions:

   Serious congenital heart disease; acute myocardial infarction within 6 months of screening; severe arrhythmias (e.g., multifocal premature ventricular tachycardia); large pericardial effusion; severe myocarditis; or hypotension requiring pressor agents at screening.
5. Pulmonary Pathology:

   1. History of severe lung disease, including significant bronchiectasis, emphysema, or advanced interstitial lung disease (ILD) at baseline.
   2. Resting oxygen saturation (SpO2 <92%).
6. Concomitant Therapy: Requirement for long-term glucocorticoids or immunosuppressive therapy for conditions other than SLE.
7. Infections: Active infections requiring systemic treatment or uncontrollable infections (bacterial, fungal, or viral) within 1 week before screening.
8. Transplantation/GVHD: Solid organ or hematopoietic stem cell transplantation within 3 months before screening; or presence of Grade 2 or higher acute graft-versus-host disease (GVHD) within 2 weeks of screening.
9. Viral and Serological Markers:

   1. Positive HBsAg or HBcAb with detectable HBV-DNA.
   2. Positive HCV antibody with detectable HCV-RNA.
   3. Positive HIV antibody, syphilis test, or detectable CMV-DNA.
10. Other Clinical Conditions:

    1. Macrophage activation syndrome (MAS) within 1 month before screening.
    2. Vaccination with a live vaccine within 4 weeks before screening.
    3. Malignancies or other severe systemic diseases.
11. Pregnancy: Positive blood pregnancy test at screening.
12. Trial Participation: Enrollment in another clinical trial within 3 months prior to this study.
13. Investigator Discretion: Any other condition that, in the opinion of the investigator, makes the subject unsuitable for the study or puts them at undue risk.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The safety of CAR-T cells in refractory Systemic Lupus Erythematosus | 3 Months
  Incidence, type, and severity of adverse events. The grading of CRS and neurotoxicity follow the ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells, published by ASTCT in 2019. Other AEs are graded using the NCI CTCAE 5.0.

SECONDARY OUTCOMES:
The efficacy of CAR-T cells in refractory Systemic Lupus Erythematosus | 3 months
  Proportion of participants achieving an SRI-4 response at 3 months post-infusion, defined by: a ≥4-point reduction in SLEDAI-2K score; no worsening in Physician's Global Assessment (increase <0.3); and no new major organ involvement as assessed by BILAG.
LLDAS response rate. | 12 months
  LLDAS response rate, defined as the percentage of subjects who meet the following conditions simultaneously after infusion: ①SLEDAI-2K score ≤4, with no activity in major organ systems (including kidney, central nervous system, heart and lungs), no vasculitis and no fever; ② no new lupus disease activity compared with the previous assessment; ③PGA score ≤1; ④serological activity permitted; ⑤ prednisolone dose ≤7.5mg daily and well-tolerated standard maintenance doses of immunosuppressive drugs or biological agents permitted.
DORIS response rate. | 12 months
  DORIS response rate, defined as the percentage of subjects who meet the following conditions simultaneously after infusion: ① clinical SLEDAI-2K score =0; ② PGA score <0.5; ③ serological activity permitted; ④low-dose glucocorticoid (i.e. prednisolone ≤5mg daily) and well-tolerated standard maintenance doses of antimalarials, immunosuppressive drugs or biological agents permitted.
Evaluate the Pharmacokinetics parameters. | 3 months
  PK parameters: The highest concentration (Cmax) of CD19-targeted CAR-T cells expanded in peripheral blood after infusion, the time to reach the highest concentration (Tmax).
Evaluate the Pharmacodynamics parameters. | 3 months
  PD parameters: The degree of B cell depletion at various time points, the concentration levels of CAR-T-related serum cytokines.
Changes in serological biomarkers related with SLE | 12 months
  Changes in serological biomarkers, including anti-dsDNA antibodies and complement C3/C4 levels, which used for evaluating the SLEDAI score

OTHER OUTCOMES:
Immune reconstitution following MC-1-50 infusion | 6 months
  To explore the impact of MC-1-50 on immune system reconstruction, including the characterization of reconstituted B-cell subsets (Naive vs. Memory) and T-cell phenotypes.
Duration of response | 12 months
  Duration of response, defined as time from first documented response to disease progression.
Optional repeat renal biopsy ≥3 months post-infusion. | 12 months
  Optional repeat renal biopsy ≥3 months post-infusion, with assessment of activity and chronicity indices, subject to separate informed consent.
Longitudinal changes in SLEDAI-2K scores over time. | 12 months
  Scores on the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) range from 0 to 105, with higher scores indicating greater disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, MD, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mackensen A, Muller F, Mougiakakos D, Boltz S, Wilhelm A, Aigner M, Volkl S, Simon D, Kleyer A, Munoz L, Kretschmann S, Kharboutli S, Gary R, Reimann H, Rosler W, Uderhardt S, Bang H, Herrmann M, Ekici AB, Buettner C, Habenicht KM, Winkler TH, Kronke G, Schett G. Anti-CD19 CAR T cell therapy for refractory systemic lupus erythematosus. Nat Med. 2022 Oct;28(10):2124-2132. doi: 10.1038/s41591-022-02017-5. Epub 2022 Sep 15. PMID 36109639
- [Result] Anders HJ, Saxena R, Zhao MH, Parodis I, Salmon JE, Mohan C. Lupus nephritis. Nat Rev Dis Primers. 2020 Jan 23;6(1):7. doi: 10.1038/s41572-019-0141-9. PMID 31974366
- [Result] Kansal R, Richardson N, Neeli I, Khawaja S, Chamberlain D, Ghani M, Ghani QU, Balazs L, Beranova-Giorgianni S, Giorgianni F, Kochenderfer JN, Marion T, Albritton LM, Radic M. Sustained B cell depletion by CD19-targeted CAR T cells is a highly effective treatment for murine lupus. Sci Transl Med. 2019 Mar 6;11(482):eaav1648. doi: 10.1126/scitranslmed.aav1648. PMID 30842314
- [Result] Jin X, Xu Q, Pu C, Zhu K, Lu C, Jiang Y, Xiao L, Han Y, Lu L. Therapeutic efficacy of anti-CD19 CAR-T cells in a mouse model of systemic lupus erythematosus. Cell Mol Immunol. 2021 Aug;18(8):1896-1903. doi: 10.1038/s41423-020-0472-1. Epub 2020 May 29. PMID 32472023
- [Result] Mougiakakos D, Kronke G, Volkl S, Kretschmann S, Aigner M, Kharboutli S, Boltz S, Manger B, Mackensen A, Schett G. CD19-Targeted CAR T Cells in Refractory Systemic Lupus Erythematosus. N Engl J Med. 2021 Aug 5;385(6):567-569. doi: 10.1056/NEJMc2107725. No abstract available. PMID 34347960
- [Result] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Result] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994